CLINICAL TRIAL: NCT02084745
Title: Timing of Glaucoma Drainage Device Implantation With Boston Keratoprosthesis Surgery
Brief Title: Timing of Glaucoma Drainage Device With Boston Keratoprosthesis
Acronym: GDD-KPro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE13.277
Record Dates: First submitted 2014-02-27; First posted 2014-03-12 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Corneal Transplantation; Glaucoma
Keywords: Boston keratoprosthesis; Glaucoma drainage device
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants

STUDY DESIGN:
Intervention Model Description: Patients will be randomized with a 1:1 allocation into two groups. Group 1 will comprise 20 patients undergoing KPro and simultaneous GDD while group 2 will include 20 patients undergoing KPro and then GDD 6 months later. Randomization schedule will be computer generated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous implantation (Active Comparator): Simultaneous implantation of a glaucoma drainage device at the time of Boston keratoprosthesis type 1 surgery
  Interventions: Procedure: Boston keratoprosthesis type 1; Procedure: Glaucoma drainage device
- Implantation at post-Kpro at 6 months (Active Comparator): Implantation of a glaucoma drainage device 6 months after Boston keratoprosthesis type 1 surgery
  Interventions: Procedure: Boston keratoprosthesis type 1; Procedure: Glaucoma drainage device

INTERVENTIONS:
Procedure: Boston keratoprosthesis type 1 — The Boston KPro, purchased from Massachusetts Eye and Ear infirmary (Boston, MA), is implanted using the usual standard technique.
  Other Names: Boston KPro type 1
Procedure: Glaucoma drainage device — The GDD that will be used is the Ahmed implant (New World Medical, Rancho Cucamonga, CA). The Ahmed implant will be implanted using the standard technique either at the time of KPro surgery in group 1, or 6 months following KPro in group 2.
  Other Names: Ahmed Glaucoma Valve

SUMMARY:
Boston keratoprosthesis (KPro) is a piece of specialized plastic that replace sick cornea (transparent structure at the front of the eye) in patients who have failed or those who are expected to have poor results with traditional corneal transplantation. While the Kpro can offer dramatic improvement in vision, it is also associated with several complications. Glaucoma (optic nerve damage due to high pressure inside the eye) is one of the most common complications after KPro surgery and can potentially cause irreversible vision loss. The implantation of a glaucoma drainage device (GDD), a tiny tube that drains the liquid inside the eye by bypassing the natural drainage system, is an effective option to lower the eye pressure in patients with KPro. Given the frequency and potentially devastating effects of glaucoma among KPro patients, some surgeons recommend to put in a GDD as a preventative measure. However, there is no consensus on when is the best timing to perform such surgery in relation to the Boston Kpro surgery.

Hypothesis:

For patients undergoing the Boston KPro surgery, implanting a GDD simultaneously, at the time of surgery, is more efficacious than at 6 months later, in the prevention of the progression of glaucoma and in maintaining better visual functions.

Methods:

The investigators aim to recruit 40 patients over 4 years. Recruited patients will be randomly assigned to 2 groups: 1) simultaneous GDD implantation at the Boston KPro surgery, and 2) GDD implantation 6 months after the Boston KPro surgery.

Once recruited, patients will be followed before the KPro surgery, postoperative day 1, week 1, month 1, 3, 6 and 12. Standard ophthalmological exam will be performed at each visit. Additional non-invasive glaucoma tests and evaluation (visual fields and optic nerve photo) will be performed on day 1, month 1, 3, 6 and 12.

For patients assigned to group 2, a GDD will be implanted 6 months after the KPro surgery. They will have additional follow-ups on post-GDD surgery day 1, week 1 and month 1.

Results of visual acuity, visual fields, optic nerve evaluation and complications will be compared between the two groups to determine the better timing of GDD implantation.

DETAILED DESCRIPTION:
INTRODUCTION:

Glaucoma is a major problem for KPro candidates. Indeed, many diagnostic indications for KPro such as aniridia, chemical burns, trauma and repeated graft failure imply alteration of the iridocorneal angle, and consequently high intraocular pressure (IOP) and glaucoma. Accordingly, the prevalence of glaucoma before KPro surgery lies between 27% and 77%, with most studies showing a prevalence above 50%. The diagnosis and management of glaucoma is particularly challenging in the KPro population. Preoperatively, the measurement of IOP is possible through Goldmann tonometry and pneumotonometry but this measurement may be erroneous due to corneal scarring and irregularity. Furthermore, corneal opacification usually prevents visualization of the optic nerve head, and visual field assessment is not possible due to poor vision. Therefore, while glaucoma is often suspected in patients undergoing KPro, this diagnosis may be only confirmed postoperatively. While optic nerve head and visual field examination become possible following KPro surgery, the determination of IOP can only be accomplished through digital palpation. The shortcomings of this method, including its very poor inter- and intra-observer reliability, are well recognized. Because IOP reduction is the basis of glaucoma treatment, it is exceedingly difficult to manage glaucoma in the KPro population. In the face of such complexity, some KPro surgeons have suggested that Glaucoma Drainage Device (GDD) implantation could be performed during KPro surgery in all patients with marginal preoperative IOP control. With this approach, the GDD could prevent postoperative IOP rise and the need for subsequent surgical and medical intervention.

RATIONALE:

The decision to implant a GDD in a patient with pre-existing or prospective KPro must be weighed carefully. The insidious development or progression of glaucoma is the most common blinding complication of KPro implantation. Indeed, the course of glaucoma is a major determinant of KPro surgery prognosis and specifically of the visual result. On the other hand, complications associated with concomitant GDD and KPro surgeries may in themselves lead to severe and irreversible vision loss and thus, prevent the visual rehabilitation of these patients. With the increasing use of the KPro, it is important to evaluate the optimal timing of GDD implantation.

HYPOTHESIS:

For patients undergoing the Boston KPro surgery, implanting a GDD simultaneously, at the time of surgery, is more efficacious than waiting 6 months to implant a GDD, in the prevention of the progression of glaucoma and in maintaining better visual acuity and visual fields

OBJECTIVE:

1. To determine the most appropriate time to implant a GDD in order to prevent the deleterious effect of glaucomatous optic neuropathy on visual rehabilitation of patients implanted with the Boston KPro.
2. To compare the outcomes of the visual acuity, visual field and glaucomatous optic disc damage by implanting a GDD at the time of KPro surgery versus implanting GDD 6 months post-KPro surgery.

METHODS:

Design: Single blind, prospective randomized controlled trial

Study Population: The duration of the study is 5 years, 4 years to recruit and 1 year to follow each patient. Forty consecutive patients (forty eyes) will be enrolled in this study. One eye of each patient will be included. The study protocol is approved by the Ethics Committee of CHUM. All patients will be informed about the design of the study and the procedure, and written informed consent will be obtained from all patients. Patient's eligibility for the study will be evaluated at the first consultation visit.

At the baseline study visit, patients will be randomized with a 1:1 allocation into two groups. Group 1 will comprise 20 patients undergoing KPro and simultaneous GDD while group 2 will include 20 patients undergoing KPro and then GDD 6 months later. Randomization schedule will be computer generated.

Prior to the surgery, a complete medical and ophthalmological history will be obtained from each patient. Patients will undergo a thorough ophthalmological evaluation, A-scan and B-scan ultrasound. The primary and concomitant pre-operative diagnoses are noted. The Boston KPro, purchased from Massachusetts Eye and Ear infirmary (Boston, MA), is implanted using the usual standard technique. The GDD that will be used is the Ahmed implant (New World Medical, Rancho Cucamonga, CA). The Ahmed implant will be implanted using the standard technique either at the time of KPro surgery in group 1, or 6 months following KPro in group 2. Standard postoperative management will be followed. Follow-up visits will be performed on day 1, week 1, and months 1, 3, 6, and 12.

Study Procedures

1. Visual acuity will be measured pre-operatively and at each visit.
2. Humphrey Visual Field 24-2 (SITA-Fast) will be performed at post-op 1 month, 3 months, 6 months, and 1 year. In cases where an automated visual field test is unreliable due to unacceptable number of false positives (>33%), false negatives (>33%), or fixation losses (>20%), a Goldmann Visual Field will be performed.
3. Optic disc examination will be done by a glaucoma specialist on post-operative days 1 and post-operative months 1, 3, 6, and 12 and graded according to the Disc Damage Likelihood Scale (DDLS). The chart containing measures of DDLS made on previous visits will not be made available to the clinician.
4. Stereoscopic photographs of the optic disc will be taken on postoperative months 1, 3, 6, 12. The blinded glaucoma specialist will assign a DDLS to each photograph.

Each patient's test results will be compiled in a table. Based on data available one month post-operatively, the investigators will decide whether there is evidence of glaucomatous optic neuropathy at this time (thereby likely reflecting presence of pre-existing glaucoma). Based on data gathered over 12 months, the investigators will decide whether or not the glaucoma has progressed through the course of the study.

All medical records, including operative protocol and progress notes, will be analyzed and data will be collected with respect to ophthalmic diagnosis of the operated eye. Patient demographics (age and gender), preoperative diagnosis, presence of pre-KPro glaucoma, surgical feasibility, retention of both GDD and KPro devices, short and long term complications of eyes who receive GDD will be studied. Patients who experience vision loss secondary to GDD complications such as tube occlusion, overfiltration, hypotony and choroidal hemorrhage will be analyzed in greater detail. Complications related to post-operative glaucoma will be evaluated. The extent of visual recuperation and the impact of glaucomatous optic nerve damage on the visual potential will be studied. Continued progression of glaucoma and the need for medical and surgical therapy will be determined.

STATISTICAL ANALYSIS:

The primary outcomes of this study, Visual Fields (Sita 24-2) and glaucomatous disc damage will be compared between both groups. Log rank test will be used to check the significance of differences between both groups. Pre- and post-best-corrected visual acuity (BCVA), as expressed in logMar units, will be compared in each group and plotted to demonstrate the evolution over time of the visual acuity in each group. Percentages of patients with fixation loss (BCVA worse than 1.30 logMar) at final visits from the two groups will also be compared.

The suitable time of GDD implantation will be determined by analyzing the visual outcome at the start and 1, 3, 6 and 12 months post-KPro and calculating the hazard on each time point. For this, time varying survival models - Cox and accelerated failure time (AFT) models will be applied according to their validity. The risk in both groups can be shown graphically by Kaplan Meier survival curve for loss of visual field and glaucomatous optic disc damage. Tests for statistical significance will be carried out at alpha=0.05.

SIGNIFICANCE:

The Boston KPro allows recovery of sight to patients with reversible corneal blindness. Glaucoma, a serious and sight threatening complication of KPro, may rob patients irreversibly and permanently of the sight they had recovered. The results of study will shed light on the most appropriate timing of glaucoma prevention and treatment. Hence, glaucoma will be treated in a timely fashion, preventing irreversible visual loss without subjecting patients to undue complications of glaucoma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for corneal transplantation due to loss of corneal clarity
* Verifiable history of one or more previous full thickness donor corneal transplantation failure
* Pre-operative visual acuity of ≤20/80 or worse in the surgical eye
* Age ≥18 years
* Physical condition suitable for undergoing surgery

Exclusion Criteria:

* Terminal glaucoma
* Terminal retinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual field mean deviation | Change from baseline visual field mean deviation at 12 months
  Humphrey Visual Field 24-2 (SITA-Fast) (or Goldmann if poor vision/reliability)

SECONDARY OUTCOMES:
Disc Damage Likelihood Scale (DDLS) on clinical examination | Change from baseline DDLS on clinical examination at 12 months
  Evaluation by a glaucoma specialist using the slit-lamp apparatus.
Disc Damage Likelihood Scale (DDLS) on stereoscopic photographs of the optic nerve | Change from baseline DDLS on optic nerve photographs at 12 months
  Outcome assessed by a glaucoma specialist blinded to previous DDLS score
Incidence of ocular complications | 12 months after KPro
  All ocular complications reported by post-KPro 12 months
Change of visual acuity | 12 months after KPro
  Change of visual acuity compared between before and after surgery. The visual acuity is measured using the Snellen chart and expressed in logMAR.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Harissi-Dagher, MD, FRCSC, Principal Investigator — Department of Ophthalmology, Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chew HF, Ayres BD, Hammersmith KM, Rapuano CJ, Laibson PR, Myers JS, Jin YP, Cohen EJ. Boston keratoprosthesis outcomes and complications. Cornea. 2009 Oct;28(9):989-96. doi: 10.1097/ICO.0b013e3181a186dc. PMID 19724214
- [Background] Banitt M. Evaluation and management of glaucoma after keratoprosthesis. Curr Opin Ophthalmol. 2011 Mar;22(2):133-6. doi: 10.1097/ICU.0b013e328343723d. PMID 21191292
- [Background] Aldave AJ, Kamal KM, Vo RC, Yu F. The Boston type I keratoprosthesis: improving outcomes and expanding indications. Ophthalmology. 2009 Apr;116(4):640-51. doi: 10.1016/j.ophtha.2008.12.058. Epub 2009 Feb 25. PMID 19243830
- [Background] Talajic JC, Agoumi Y, Gagne S, Moussally K, Harissi-Dagher M. Prevalence, progression, and impact of glaucoma on vision after Boston type 1 keratoprosthesis surgery. Am J Ophthalmol. 2012 Feb;153(2):267-274.e1. doi: 10.1016/j.ajo.2011.07.022. Epub 2011 Oct 7. PMID 21982110